CLINICAL TRIAL: NCT01301989
Title: Reducing Sleep Disparities in Urban, Minority School-Aged Children
Brief Title: Reducing Sleep Disparities in Minority Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Beverley J Sheares MD, MS, Assoc Professor of Pediatrics at CUMC, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAE4951; R01HL092856 (NIH)
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Sleep
Keywords: Sleep; Children; Disparities; Minority; Urban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep Education Control (Placebo Comparator): The control group receives a low intensity intervention that provides information about sleep and the benefits of adequate sleep. We will give parents the National Sleep Foundation's handout, "Information about Children's Sleep for Parents and Teachers" (in English and Spanish).
  Interventions: Other: Sleep Education Control
- Sleep Counselor Intervention (Experimental): The sleep counselor visits are to assess the family's understanding of their child's sleep problems; help parents recognize the child's sleep deficiency; discuss how sleep problems affect behavior, learning, and health; and reassure parents that the sleep counselor can help them with these problems.
  Additionally, sleep counselors: review parent's sleep goals to monitor changes to the child's bedtime routine and sleep environment; help them solve problems with implementation; provide positive feedback to help the parent recognize success; and help parents set additional goals for improving sleep.
  Interventions: Behavioral: Sleep Counselor Intervention

INTERVENTIONS:
Behavioral: Sleep Counselor Intervention — Families in the sleep counselor arm of the study will receive 3 scheduled home visits by a trained sleep counselor during the first 3 months following enrollment. Two optional home visits may be scheduled to help families encountering ongoing barriers to improving their child's sleep. The intervention will be provided by trained, bilingual, culturally competent sleep counselors, who will assess home sleep conditions, work with the family to teach them how to improve sleep hygiene and the sleep environment, provide equipment as needed to improve the sleep environment (e.g. nightlight, inflatable bed, window shade, etc.) and guide the family to begin setting goals and making decisions to initiate and sustain behavioral and environmental changes to improve sleep.
  Arms: Sleep Counselor Intervention
Other: Sleep Education Control — The control group will receive a low intensity intervention that provides information about sleep and the benefits of adequate sleep. We will give parents the National Sleep Foundation's handout, "Information about Children's Sleep for Parents and Teachers"
  Arms: Sleep Education Control

SUMMARY:
Inadequate sleep is a major health problem of childhood that often fails to receive attention until significant neurobehavioral and other health problems are noted. Although adequate sleep is essential for normal growth and brain development, studies show that children from minority and economically disadvantaged families are more likely to experience shorter sleep times and more sleep fragmentation compared to their Caucasian and economically advantaged counterparts. As a result, they are disproportionately affected by the adverse health and quality of life consequences of poor sleep. There are currently no intervention studies to the investigators knowledge aimed at addressing sleep disparities by improving sleep duration and sleep hygiene in early school-aged children from minority populations. This study seeks to close the 'sleep gap' that exists between the sleep duration of minority school-aged children and that of their non-minority peers. An interdisciplinary team of researchers and clinicians from Columbia University's Pediatric Lung and Sleep Disorders Center, School of Public Health, Psychiatry Department, and two outpatient clinic systems affiliated with Columbia are collaborating to reduce sleep disparities by improving sleep duration in a group of 5-6 year old minority children. The primary goal of this study is to evaluate the efficacy of a tailored, interactive, educational and behavioral intervention that utilizes trained sleep counselors to assist parents in improving their children's sleep hygiene and reducing risk factors for poor sleep, thereby increasing sleep duration over a 12-month period in a randomized controlled trial of children identified with sleep problems (Aim 1). The investigators will screen 375 parents of 5-6 year old children from 5 primary care clinics to identify children with and without sleep problems and enroll 90 of the 375 children screened who have sleep problems in a randomized controlled trial of an in-home sleep intervention. Using an initial home assessment, baseline actigraphy data, sleep logs recorded by parents, and information regarding risk factors for poor sleep collected from each family during screening, the investigators will work with intervention parents to develop a personalized sleep plan for their children. The investigators will evaluate the effect of the intervention on: a) nightly sleep duration; b) neurocognitive function; and c) behavioral disorders.

DETAILED DESCRIPTION:
Inclusion Criteria. Eligible families must: (1) have a typically developing healthy child age 5-6 years old enrolled in school for a minimum of 5 hours per day; (2) have a child who screens positive for a sleep problem based on the CSHQ (a score >41); (3) have lived in permanent housing within the catchment communities for the study (not in a shelter or other temporary housing) for the previous 12 months; (4) have no plans to move out of the area in the next 12 months; (5) agree to have research staff come into their homes for a home assessment and actigraph fitting every 3 months for 1 year; (6) have telephone access or a contact with telephone access; and (7) be fluent in either English or Spanish.

Exclusion criteria will include the presence of a serious co-morbid condition in the child that may impact sleep including: genetic syndromes, neuromuscular disorders, seizure disorder, mental retardation, autism, severe learning disabilities, psychiatric disorders, and attention-deficit/hyperactivity disorder. The presence of such co-morbid conditions would confound the outcome of interest.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child age 5-6 years old
* School enrollment for a minimum of 5 hours/day
* Positive Children's Sleep Habits Questionnaire (score ≥ 41)
* Permanent housing for the previous 12 months
* Permission for research staff to complete 5-9 home over 1 year
* Have telephone access or a contact with telephone access
* Fluent in either English or Spanish

Exclusion Criteria:

* Serious co-morbid condition that may impact sleep including:

  * genetic syndromes
  * neuromuscular disorders
  * seizure disorder
  * mental retardation
  * autism
  * severe learning disabilities
  * psychiatric disorders
  * attention-deficit/hyperactivity disorder

Ages: 60 Months to 87 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sleep Duration | Baseline and 3 month intervals for 12 months
  The primary outcome is nightly sleep duration and is objectively measured using actigraphy. The actigraph is worn on the non-dominant wrist for 7 consecutive days and nights. Actigraphy is a well-validated method for evaluating sleep and circadian rhythm patterns in children. It is highly correlated with polysomnography. To reduce potential confounders, Actiwatches are worn 5 times during the study, at baseline and at 3, 6, 9, 12 months following collection of baseline data.

SECONDARY OUTCOMES:
Sleep Fragmentation | Baseline, 3, 6, 9, and 12 months
  Sleep fragmentation (average number and duration of nightly awakenings in each 7-day period) measured by actigraphy and parental sleep logs.

CONTACTS AND LOCATIONS:
Overall Officials: Beverley J Sheares, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Sheares BJ, Kattan M, Leu CS, Lamm CI, Dorsey KB, Evans D. Sleep problems in urban, minority, early-school-aged children more prevalent than previously recognized. Clin Pediatr (Phila). 2013 Apr;52(4):302-9. doi: 10.1177/0009922813476573. Epub 2013 Feb 19. PMID 23426232